CLINICAL TRIAL: NCT02558972
Title: Northera Improves Postural Tachycardia Syndrome (POTS) and Postural
Brief Title: Northera Improves Postural Tachycardia Syndrome (POTS) and Postural Vasovagal Syncope (VVS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not recruit adequate numbers. Largely closed by COVID risk.
Sponsor: New York Medical College (Other)
Collaborators: Lundbeck LLC (Industry)
Responsible Party: Principal Investigator, Julian Stewart, Professor of Pediatrics and Physiology, New York Medical College
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L-11,388
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Postural Tachycardia Syndrome (POTS); Vasovagal Syncope (VVS); Fainting
Keywords: Postural Tachycardia Syndrome (POTS); Vasovagal Syncope (VVS); Fainting; Orthostatic Intolerance; Droxidopa; Northera
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Syncope, Vasovagal; Syncope; Orthostatic Intolerance | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Northera-single dose (Placebo Comparator): Study #1 -Does single large dose (600mg) of Northera improve upright hemodynamics and orthostatic intolerance in POTS and VVS
  Interventions: Drug: Northera (Droxidopa); Drug: Placebo
- Northera- chronic administration (Placebo Comparator): Study #2 -Patients will randomized to receive Northera or placebo for two weeks after which they will return for instrumented tilt studies as in Study 1. Doses of Northera will be titrated upwards by 100mg/dose every 48 hours from a starting dose of 100mg three times a day to a maximum of 600mg three times a day.
  Interventions: Drug: Northera (Droxidopa); Drug: Placebo

INTERVENTIONS:
Drug: Northera (Droxidopa) — Study #1 -Supine monitoring is performed for 30 minutes before administration of a single 600mg oral dose of Northera or placebo assigned randomly, After 2 hours supine a 70 degree upright tilt will performed for 10 minutes. On another day, subjects previously given Northera will receive placebo and vice versa and studies repeated.
  Arms: Northera-single dose
Drug: Placebo — Study #1 -Supine monitoring is performed for 30 minutes before administration of a single 600mg oral dose of Northera or placebo assigned randomly, After 2 hours supine a 70 degree upright tilt will performed for 10 minutes. On another day, subjects previously given Northera will receive placebo and vice versa and studies repeated.
  Arms: Northera-single dose
Drug: Northera (Droxidopa) — Study #2 -Patients will randomized to receive Northera or placebo for two weeks after which they will return for instrumented tilt studies as in Study 1. Doses of Northera will be titrated upwards by 100mg/dose every 48 hours from a starting dose of 100mg three times a day to a maximum of 600mg three times a day. Doses will be reduced to the preceding dose if systolic BP>140mmHg or diastolic BP>80mmHg measured in the seated position at home using an automated ambulatory blood pressure cuff 2 hours after receiving an oral dose. Doses will also be reduced if supine BP measured with the head of the bed elevated upon awakening in the morning exceeds 150/90 mmHg. Following a 1 week wash out period, subjects will receive the alternative treatment for 2 additional weeks and instrumented laboratory studies repeated.
  Arms: Northera- chronic administration
Drug: Placebo — Study #2 -Patients will randomized to receive Northera or placebo for two weeks after which they will return for instrumented tilt studies as in Study 1. Doses of Northera will be titrated upwards by 100mg/dose every 48 hours from a starting dose of 100mg three times a day to a maximum of 600mg three times a day. Doses will be reduced to the preceding dose if systolic BP>140mmHg or diastolic BP>80mmHg measured in the seated position at home using an automated ambulatory blood pressure cuff 2 hours after receiving an oral dose. Doses will also be reduced if supine BP measured with the head of the bed elevated upon awakening in the morning exceeds 150/90 mmHg. Following a 1 week wash out period, subjects will receive the alternative treatment for 2 additional weeks and instrumented laboratory studies repeated.
  Arms: Northera- chronic administration

SUMMARY:
Vasovagal syncope (VVS, simple faint) is the most common cause of transient loss of consciousness and represents the acute episodic form of orthostatic intolerance (OI). Postural tachycardia syndrome (POTS) is the common chronic form of OI. Both are defined by debilitating symptoms and signs while upright relieved by recumbency. Northera should therefore improve both sympathetic splanchnic arterial vasoconstriction and sympathetic splanchnic venoconstriction in POTS and VVS, and may represent an ideal drug to improve the orthostatic response in POTS and VVS.

DETAILED DESCRIPTION:
Vasovagal syncope (VVS, simple faint) is the most common cause of transient loss of consciousness and represents the acute episodic form of orthostatic intolerance (OI). Postural tachycardia syndrome (POTS) is the common chronic form of OI. Both are defined by debilitating symptoms and signs while upright relieved by recumbency. Pathophysiological mechanisms have remained elusive. Most POTS patients and all VVS patients have normal supine resting hemodynamics but excessively redistribute blood flow and blood volume from the central pool to the splanchnic vasculature because of defective splanchnic arterial vasoconstriction and venoconstriction. While peripheral and splanchnic arterial vasoconstriction depend primarily on post-junctional alpha-1 adrenergic receptors, splanchnic venoconstriction also depends on post-junctional alpha-2 adrenergic receptors. Consequently, selective alpha-1 agonists such as midodrine may not produce sufficient splanchnic venoconstriction to compensate for splanchnic pooling in POTS and VVS. Such alpha adrenergic subtype restrictions do not apply to Northera (droxidopa) because it is a norepinephrine (NE) prodrug and therefore increases the amount of synaptic NE that can then bind to both alpha-2 and alpha-1 receptors. Northera should therefore improve both sympathetic splanchnic arterial vasoconstriction and sympathetic splanchnic venoconstriction in POTS and VVS, and may represent an ideal drug to improve the orthostatic response in POTS and VVS. We will test the hypothesis that Northera, in appropriate dose, improves the splanchnic adrenergic deficits that initiate POTS and postural VVS and in sufficient daily dose improves quality of life in these patients. To accomplish this, the investigator will recruit 10 POTS patients aged 18-30 years, 10 similarly aged patients with 2 or more episodes of VVS in the past year (thus defining recurrent VVS) and 10 age and gender matched healthy volunteer control subjects with the following specific aims:

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants are being studied
* Ages 18-30 years old
* POTS cases will be referred for day-to-day Orthostatic Intolerance (OI) with ≥3 symptoms for >6 months.
* POTS will be confirmed by medical history indicating chronic OI, and by a prior 700 tilt table test or standing test showing excessive tachycardia and symptoms OI in the absence of hypotension.
* VVS (fainting) subjects will have at least 2 episodes of postural VVS during the past calendar year.
* Healthy volunteers will be included for Study #1

Exclusion Criteria:

* Only those free from all systemic illnesses will be eligible to participate. This excludes patients with illnesses associated with autonomic dysfunction such as diabetes, renal disease, congestive heart failure, systemic hypertension, acute and chronic inflammatory diseases, neoplasm, immune mediated disease, trauma, obesity, cancer, supine or upright hypertension, and peripheral vascular disease.
* No subjects will be taking neurally active, or vasoactive drugs. Prior medication will be stopped for at least 2 weeks.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Study #1 and Study #2 - Splanchnic and lower extremity pooling (physiological parameter) | 2 weeks
  Splanchnic and lower extremity pooling will be measured before, during, and after upright tilt. The investigators will use both venous occlusion plethysmography and impedance plethysmography. Venous occlusion plethysmography are made in ml/min by rapidly inflating cuffs to a pressure of 45mmHg and then computing the slope of the time dependent increase in cross limb section. During impedance plethysmography, a Tetrapolar High Resolution Impedance monitor 4-channel digital IPG is used to detect changes in regional blood volume and blood flow in ml/min
Study #2 -Quality of Life measured by self reporting questionnaire (RAND-36) | 6 weeks
  The investigators will test whether chronic administration of Northera (Droxidopa) in escalating dose improves quality of life. Quality of life will be measured by the RAND-36 questionnaire. The RAND-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. (2-4)
Study #2 -Quality of Life measured by self reporting questionnaire (COMPASS 31) | 6 weeks
  The investigators will test whether chronic administration of Northera (Droxidopa) in escalating dose improves quality of life. Quality of life will be measured by the RAND-36 questionnaire (as shown in the above primary outcome) as well as the COMPASS 31 questionnaire. The COMPASS 31 "was developed as a self-assessment instrument of autonomic symptoms and function that is up-to-date, broadly applicable, easy to administer in a short amount of time, and based on a scientific approach. It was designed to provide a global autonomic severity score and domain scores that are both clinically and scientifically meaningful." "COMPASS 31 is based on the well-established ASP [Autonomic Symptom Profile], a comprehensive questionnaire assessing autonomic symptoms across multiple domains." (1)

SECONDARY OUTCOMES:
Study #1 and Study #2 -Blood pressure (BP) | 2 weeks
  During laboratory testing, blood pressure will be continuously monitored in mmHg
Study #1 and Study #2 -Heart rate (HR) | 2 weeks
  During laboratory testing, heart rate will be continuously monitored in beats/minute.

CONTACTS AND LOCATIONS:
Overall Officials: Julian M Stewart, M.D., Ph.D., Principal Investigator — New York Medical College
Locations (1):
- New York Medical College/Bradhurst building, Hawthorne, New York, United States

REFERENCES:
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] http: and www.rand.org/health/surveys_tools/mos/mos_core_36item.html. 36-Item Short Form Survey from the RAND Medical Outcomes Study. 2014.
- [Background] Hays RD, Shapiro MF. An overview of generic health-related quality of life measures for HIV research. Qual Life Res. 1992 Apr;1(2):91-7. doi: 10.1007/BF00439716. PMID 1301123
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- See also: The Center for Hypotension — http://syncope.org